CLINICAL TRIAL: NCT02191085
Title: Evaluation of a "Fast Track" Respiratory Therapy Clinic for Patients With Suspected Severe Sleep-Disordered Breathing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: The Lung Association (Unknown)
Responsible Party: Principal Investigator, Sachin R. Pendharkar, Dr., University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: REB13-1280
Record Dates: First submitted 2014-07-13; First posted 2014-07-15 (Estimated); Results first posted 2025-07-10 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Sleep Disordered Breathing
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Management (No Intervention): Patients in the "Standard Management" arm will be assessed without any interventions.Patients will be assessed by a sleep respirologist and follow a management plan that is determined by the sleep physician and patient. This plan may involve polysomnography or the initiation of PAP therapy. If further testing is ordered, follow-up may occur with the physician or with an ACP, at the physician's discretion. For patients initiating PAP therapy, the decision to delegate follow-up to an ACP will be left up to the physician, as the intent of this study is to observe real-world practice and not to change the management of individual patients.
- Fast Track (Active Comparator): In the "Fast Track" arm, an ACP will perform the initial assessment and will determine the management plan with the patient.
  Interventions: Procedure: Fast Track

INTERVENTIONS:
Procedure: Fast Track — In the "Fast Track" arm, an ACP will perform the initial assessment and will determine the management plan with the patient. To ensure patient safety, the management plan will be discussed with a sleep respirologist, who will be designated as the patient's primary sleep physician. This sleep physician will be available at the FMC Sleep Centre during the "Fast Track" clinic to assist with the assessment of patients who appear unwell. As in the "Standard Management" arm, follow-up visits to review test results, discuss and initiate treatment, or to assess treatment response may occur with the ACP who performed the initial assessment or may be delegated to any other ACP.
  Arms: Fast Track

SUMMARY:
Access to medical care for patients with breathing disorders during sleep is a major problem for Canadians. Recently, there has been increasing interest in how health care providers who are not physicians can help to improve access to medical care for these patients, but it is unclear whether patients with severe sleep-disordered breathing who receive care from these non-physician providers have the same response to treatment as patients who receive care from physicians. Since these severe have a high risk of developing cardiac and respiratory complications and of being hospitalized, an initiative to improve access such as the use of non-physician providers could be of great benefit to individual patients and the health care system.

The objectives of this project are:

1. to determine whether patients with severe breathing disorders during sleep have the same response to treatment when cared for by non-physician health care providers (respiratory therapists) as they do when cared for by physicians;
2. to determine the effects of non-physician health care provider treatment to patient access;
3. to determine health care utilization and related costs associated with non-physician health care provider treatment.

DETAILED DESCRIPTION:
The difficulty in providing timely access to sleep specialists is widespread. These delays are particularly important for patients with severe sleep-disordered breathing (SDB) due to the increased risk of adverse clinical outcomes and potential associated healthcare costs. The lack of timely access has sparked an interest in the use of alternate care providers (ACPs) to manage patients with SDB. Our group and others have demonstrated that ACPs are an effective and efficient substitute for physicians for patients with uncomplicated SDB. However, the role of ACPs in the management of patients with severe SDB remains unclear.

Prompted by wait times that far exceed current Canadian guidelines, we have recently implemented an ACP-led "Fast Track" clinic for patients who are referred to the Foothills Medical Centre (FMC) Sleep Centre with suspected severe SDB. In this clinic, patients with suspected severe SDB are assessed by a sleep-trained registered respiratory therapist functioning as an ACP. Decisions regarding further sleep testing and treatment are made by the patient and ACP, under the guidance of a sleep physician. This model of care differs from a physician-led model that is used at the FMC Sleep Centre.

To evaluate this novel care delivery model, we have designed a randomized trial comparing outcomes for patients in the "Fast Track" clinic to those who undergo conventional, physician-led care. The specific goals of this study are:

1. to compare the clinical effectiveness of an ACP-led clinic for patients with suspected severe SDB to physician-led management;
2. to determine whether cycle times from referral to diagnosis and treatment for patients referred with suspected severe SDB can be reduced by an ACP-led clinic;
3. to determine the impact of an ACP-led clinic on the demand for sleep physicians, ACPs and diagnostic testing;
4. to compare the cost-effectiveness of these models of care using data on healthcare utilization, costs, and patient reported health-related quality of life (HRQOL).

Patients in the "Standard Management" arm will be assessed by a sleep respirologist and follow a management plan that is determined by the sleep physician and patient. This plan may involve polysomnography or the initiation of positive airway pressure (PAP) therapy. If further testing is ordered, follow-up may occur with the physician or with an ACP, at the physician's discretion. For patients initiating PAP therapy, the decision to delegate follow-up to an ACP will be left up to the physician, as the intent of this study is to observe real-world practice and not to change the management of individual patients.

In the "Fast Track" arm, an ACP will perform the initial assessment and will determine the management plan with the patient. To ensure patient safety, the management plan will be discussed with a sleep respirologist, who will be designated as the patient's primary sleep physician. This sleep physician will be available at the FMC Sleep Centre during the "Fast Track" clinic to assist with the assessment of patients who appear unwell (e.g. severe hypoxemia, decompensated cardiorespiratory failure, etc.). As in the "Standard Management" arm, follow-up visits to review test results, discuss and initiate treatment, or to assess treatment response may occur with the ACP who performed the initial assessment or may be delegated to any other ACP.

As is usual procedure at the FMC Sleep Centre, ambulatory sleep test requisitions will be completed by ACPs or physicians, whereas all polysomnogram requisitions will be completed by the primary sleep physician to ensure adequate blinding of patient assignment. The research associate will ensure that all tests are interpreted in advance of clinic visits. Patients who are followed by ACPs in either arm can be referred to the primary sleep physician for assessment of non-respiratory sleep disorders, or for persistent symptoms such as daytime sleepiness.

ELIGIBILITY:
Inclusion Criteria:

* referred to the FMC Sleep Centre for assessment of SDB
* meet one of the three criteria for suspected severe SDB:

  1. Respiratory disturbance index (RDI) >/= 30 events/hour on an ambulatory sleep test
  2. Mean nocturnal oxygen saturation </= 85% on an ambulatory sleep test
  3. Suspected hypoventilation, defined by an RDI >/= 15 events/hour on an ambulatory sleep test and partial pressure of carbon dioxide >/= 45 mmHg on arterial blood gas
  4. On supplemental oxygen therapy with high suspicion of SDB (as determined by physician review of referral)

Exclusion Criteria:

* Suspected concomitant sleep disorder other than SDB
* A previous diagnosis of OSA treated with PAP or dental appliance
* Primary health insurance provided by a province other than Alberta
* Failure to provide consent to participate in the study
* Under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sachin R Pendharkar, MD, MSc, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre Sleep Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marin JM, Carrizo SJ, Vicente E, Agusti AG. Long-term cardiovascular outcomes in men with obstructive sleep apnoea-hypopnoea with or without treatment with continuous positive airway pressure: an observational study. Lancet. 2005 Mar 19-25;365(9464):1046-53. doi: 10.1016/S0140-6736(05)71141-7. PMID 15781100
- [Background] Yaggi HK, Concato J, Kernan WN, Lichtman JH, Brass LM, Mohsenin V. Obstructive sleep apnea as a risk factor for stroke and death. N Engl J Med. 2005 Nov 10;353(19):2034-41. doi: 10.1056/NEJMoa043104. PMID 16282178
- [Background] Peppard PE, Young T, Palta M, Skatrud J. Prospective study of the association between sleep-disordered breathing and hypertension. N Engl J Med. 2000 May 11;342(19):1378-84. doi: 10.1056/NEJM200005113421901. PMID 10805822
- [Background] Flemons WW, Tsai W. Quality of life consequences of sleep-disordered breathing. J Allergy Clin Immunol. 1997 Feb;99(2):S750-6. doi: 10.1016/s0091-6749(97)70123-4. PMID 9042067
- [Background] Reimer MA, Flemons WW. Quality of life in sleep disorders. Sleep Med Rev. 2003 Aug;7(4):335-49. doi: 10.1053/smrv.2001.0220. PMID 14505600
- [Background] Berg G, Delaive K, Manfreda J, Walld R, Kryger MH. The use of health-care resources in obesity-hypoventilation syndrome. Chest. 2001 Aug;120(2):377-83. doi: 10.1378/chest.120.2.377. PMID 11502632
- [Background] Redline S, Yenokyan G, Gottlieb DJ, Shahar E, O'Connor GT, Resnick HE, Diener-West M, Sanders MH, Wolf PA, Geraghty EM, Ali T, Lebowitz M, Punjabi NM. Obstructive sleep apnea-hypopnea and incident stroke: the sleep heart health study. Am J Respir Crit Care Med. 2010 Jul 15;182(2):269-77. doi: 10.1164/rccm.200911-1746OC. Epub 2010 Mar 25. PMID 20339144
- [Background] Antic NA, Buchan C, Esterman A, Hensley M, Naughton MT, Rowland S, Williamson B, Windler S, Eckermann S, McEvoy RD. A randomized controlled trial of nurse-led care for symptomatic moderate-severe obstructive sleep apnea. Am J Respir Crit Care Med. 2009 Mar 15;179(6):501-8. doi: 10.1164/rccm.200810-1558OC. Epub 2009 Jan 8. PMID 19136368
- [Derived] J Santana M, Jaja O, Duan Q, D Penz E, L Fraser K, J Hanly P, R Pendharkar S. Comparison of patient-reported outcomes between alternative care provider-led and physician-led care for severe sleep disordered breathing: secondary analysis of a randomized clinical trial. J Patient Rep Outcomes. 2024 Sep 26;8(1):107. doi: 10.1186/s41687-024-00747-3. PMID 39325310
- [Derived] Thornton CS, Tsai WH, Santana MJ, Penz ED, Flemons WW, Fraser KL, Hanly PJ, Pendharkar SR. Effects of Wait Times on Treatment Adherence and Clinical Outcomes in Patients With Severe Sleep-Disordered Breathing: A Secondary Analysis of a Noninferiority Randomized Clinical Trial. JAMA Netw Open. 2020 Apr 1;3(4):e203088. doi: 10.1001/jamanetworkopen.2020.3088. PMID 32310283
- [Derived] Pendharkar SR, Tsai WH, Penz ED, Santana MJ, Ip-Buting A, Kelly J, Flemons WW, Fraser KL, Hanly PJ. A Randomized Controlled Trial of an Alternative Care Provider Clinic for Severe Sleep-disordered Breathing. Ann Am Thorac Soc. 2019 Dec;16(12):1558-1566. doi: 10.1513/AnnalsATS.201901-087OC. PMID 31437008
- [Derived] Ip-Buting A, Kelly J, Santana MJ, Penz ED, Flemons WW, Tsai WH, Fraser KL, Hanly PJ, Pendharkar SR. Evaluation of an alternative care provider clinic for severe sleep-disordered breathing: a study protocol for a randomised controlled trial. BMJ Open. 2017 Mar 29;7(3):e014012. doi: 10.1136/bmjopen-2016-014012. PMID 28360244

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Management | Fast Track
Started | 92 | 94
Included in Modified Intention to Treat Population | 75 | 81
Completed | 75 (Received allocated intervention) | 81 (Received allocated intervention)
Not Completed | 17 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Management | Fast Track | Total
Number analyzed (Participants) | 92 | 94 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Reported number reflects those that received intervention as per modified intention to treat design
  years
    number analyzed (Participants) | 75 | 81 | 156
    (all) | 55 (13) | 54 (12) | 55 (12)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Reported number reflects those that received intervention as per modified intention to treat design
  Participants
    number analyzed (Participants) | 75 | 81 | 156
    Female | 21 | 23 | 44
    Male | 54 | 58 | 112
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 92 | 94 | 186
Body mass index, kg/m^2 [Mean (Standard Deviation); unit: kg/m^2] — Population: Reported number reflects those that received intervention as per modified intention to treat design
  kg/m^2
    number analyzed (Participants) | 75 | 81 | 156
    (all) | 39 (9) | 40 (10) | 39 (10)
Respiratory Event Index, events/h [Mean (Standard Deviation); unit: events/h] — Respiratory Event Index on level 3 home sleep apnea test, collected at baseline Population: Reported number reflects those that received intervention as per modified intention to treat design
  events/h
    number analyzed (Participants) | 75 | 81 | 156
    (all) | 55 (29) | 51 (28) | 53 (28)
Mean oxygen saturation on home sleep apnea test [Mean (Standard Deviation); unit: % oxygen saturation] — Mean oxygen saturation during a level 3 home sleep apnea test, collected at baseline Population: Reported number reflects those that received intervention as per modified intention to treat design
  % oxygen saturation
    number analyzed (Participants) | 75 | 81 | 156
    (all) | 86 (5) | 85 (5) | 85 (5)
Apnea hypopnea index, events/h [Mean (Standard Deviation); unit: events/h] — Apnea hypopnea index measured using level 1 polysomnography, measured to characterize sleep-disordered breathing in selected patients. Need for polysomnography was determined by the clinical provider at initial assessment. This measurement was not performed at baseline but was not influenced by study allocation and is provided as another baseline measure of sleep-disordered breathing severity. Population: Reported number reflects those that received intervention as per modified intention to treat design and who underwent polysomnography
  events/h
    number analyzed (Participants) | 46 | 40 | 86
    (all) | 77 (50) | 75 (59) | 76 (54)
Mean oxygen saturation on polysomnography [Mean (Standard Deviation); unit: % oxygen saturation] — Mean oxygen saturation measured during level 1 polysomnography, measured to characterize sleep-disordered breathing in selected patients. Need for polysomnography was determined by the clinical provider at initial assessment. This measurement was not performed at baseline but was not influenced by study allocation and is provided as another baseline measure of sleep-disordered breathing severity. Population: Reported number reflects those that received intervention as per modified intention to treat design and who underwent polysomnography
  % oxygen saturation
    number analyzed (Participants) | 46 | 40 | 86
    (all) | 86 (5) | 85 (5) | 85 (5)

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Positive Airway Pressure (PAP) Therapy
Description: Data includes number of hours used per night on all nights
Time Frame: 3 months after treatment initiation
Measure: Mean (95% Confidence Interval); unit: hours per night
Arm/Group | Standard Management | Fast Track
Number analyzed (Participants) | 75 | 81
hours per night | 4 [3.3 to 4.7] | 3.5 [2.8 to 4.2]

2. Secondary Outcome: Change in Daytime Sleepiness
Description: Epworth Sleepiness Scale - this is a subjective scale measuring tendency for an individual to fall asleep in 8 different circumstances. Score is 0-3 for each circumstance but is reported as a total score.
  Minimum total score = 0, Maximum total score = 24 Higher scores mean worse outcome
Time Frame: 3 months after treatment initiation
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Standard Management | Fast Track
Number analyzed (Participants) | 60 | 67
score on a scale | 3.4 [1.8 to 5] | 5.4 [4.3 to 6.8]

3. Secondary Outcome: Health Care Utilization
Description: Costs for physician visits, emergency department visits, hospitalizations
Time Frame: 1 year after treatment initiation
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Standard Management | Fast Track
Number analyzed (Participants) | 75 | 81
dollars
  Physician costs | 1960 (2440) | 1670 (2430)
  Emergency Department visits | 282 (831) | 219 (585)
  Hospitalization visits | 1410 (4410) | 1760 (5930)

4. Secondary Outcome: Total Healthcare Costs
Description: Comparing costs for each arm (used to calculate the incremental cost effectiveness ratio)
Time Frame: 1 year after treatment initiation
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Standard Management | Fast Track
Number analyzed (Participants) | 75 | 80
dollars | 8572 (7617) | 8203 (8841)

5. Secondary Outcome: Time From Date of Referral to Date of Treatment Initiation
Description: Comparing cycle times for intervention vs. control arm
Time Frame: Expected within 1 year (unknown due to nature of outcome)
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Standard Management | Fast Track
Number analyzed (Participants) | 75 | 81
days | 134 [121 to 147] | 110 [94 to 125]

6. Secondary Outcome: Change in Daytime Sleepiness
Description: Epworth Sleepiness Scale - a subjective scale measuring tendency for an individual to fall asleep in 8 different circumstances. Total score is sum of score in each circumstance (0-3) Minimum total score = 0, Maximum total score = 24 Higher scores mean worse outcome
Time Frame: 1 year after treatment initiation
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Management | Fast Track
Number analyzed (Participants) | 37 | 44
units on a scale | 4.62 [2.37 to 6.88] | 1.79 [0.97 to 4.55]

7. Secondary Outcome: Adherence to Positive Airway Pressure (PAP) Therapy
Description: Data includes number of hours used per night.
Time Frame: 1 year after treatment initiation
Measure: Mean (95% Confidence Interval); unit: hours/night
Arm/Group | Standard Management | Fast Track
Number analyzed (Participants) | 37 | 38
hours/night | 5.56 [4.76 to 6.35] | 6.14 [5.44 to 6.85]

8. Secondary Outcome: Change in Disease Specific Health-related Quality of Life
Description: Sleep Apnea Quality of Life Index - subjective disease-specific quality of life scale, incorporating 4 domains measured pre/post intervention (scored 1-7 on a Likert scale) and 3 post-intervention domains that are weighted before incorporated in the final score Minimum = 1 Maximum = 7 Higher scores indicate a better outcome
Time Frame: 3 months after treatment initiation
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Management | Fast Track
Number analyzed (Participants) | 60 | 66
units on a scale | 0.83 [0.5 to 1.2] | 1.2 [0.9 to 1.5]

9. Secondary Outcome: Change in Disease Specific Health-related Quality of Life
Description: as for outcome 8
Time Frame: 1 year after treatment initiation
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Management | Fast Track
Number analyzed (Participants) | 37 | 44
units on a scale | 0.99 [0.45 to 1.53] | 1.39 [1 to 1.78]

10. Secondary Outcome: Patient Satisfaction
Description: Visit-Specific Instrument (VSQ-9) - comprises 9 questions for which patients assign a Likert scale score from 0-5. Score is reported as sum of Likert scale score for each question 0 to 45 scale Higher scores mean a better outcome.
Time Frame: 3 months after treatment initiation
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Management | Fast Track
Number analyzed (Participants) | 50 | 56
units on a scale | 36 [34 to 38] | 38 [36 to 39]

11. Secondary Outcome: Patient Satisfaction
Description: as for outcome 10
Time Frame: 1 year after treatment initiation
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Management | Fast Track
Number analyzed (Participants) | 35 | 44
units on a scale | 34.54 [31.74 to 37.34] | 37.39 [35.54 to 39.23]

12. Secondary Outcome: Number of Sleep Diagnostic Tests and Sleep Ambulatory Care Visits
Description: Reported as costs for home sleep apnea tests, polysomnograms, new and follow-up clinical visits
Time Frame: 1 year after treatment initiation
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Standard Management | Fast Track
Number analyzed (Participants) | 75 | 81
dollars
  Home sleep apnea test costs | 57.2 (21.4) | 56.2 (20.3)
  Polysomnogram costs | 649 (589) | 566 (637)
  New clinical visit costs | 182 (0) | 56.2 (0)
  Follow-up clinical visits | 101 (119) | 77.6 (91.3)

13. Secondary Outcome: Change in Severity of Sleep-disordered Breathing
Description: Respiratory event index from ambulatory testing - reported values represent change from baseline to 3 months
Time Frame: baseline and 3 months after treatment initiation
Measure: Mean (95% Confidence Interval); unit: events/h
Arm/Group | Standard Management | Fast Track
Number analyzed (Participants) | 55 | 61
events/h | -45 [-53 to -38] | -41 [-48 to -34]

14. Secondary Outcome: Change in Severity of Sleep-disordered Breathing
Description: Respiratory event index from ambulatory testing - reported values represent change from baseline to 3 months
Time Frame: baseline and 1 year after treatment initiation
Measure: Mean (95% Confidence Interval); unit: events/h
Arm/Group | Standard Management | Fast Track
Number analyzed (Participants) | 33 | 32
events/h | -46 [-58 to -33] | -44 [-56 to -32]

15. Secondary Outcome: Change in General Health-related Quality of Life
Description: Health Utilities Index - a 17-question general health related quality of life index. Total score indicates subjective assessment of HRQOL from close to death to perfect health Maximum = 1 Minimum = 0 Higher score means a better outcome
Time Frame: 3 months after treatment initiation
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Management | Fast Track
Number analyzed (Participants) | 60 | 66
units on a scale | 0.06 [-0.01 to 0.14] | 0.15 [0.08 to 0.21]

16. Secondary Outcome: Change in General Health-related Quality of Life
Description: as for outcome 15
Time Frame: 1 year after treatment initiation
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Management | Fast Track
Number analyzed (Participants) | 37 | 44
units on a scale | 0.15 [0.05 to 0.24] | 0.15 [0.06 to 0.23]

17. Secondary Outcome: Quality Adjusted Life Years
Description: Comparing quality adjusted life years for each arm (used to calculate the incremental cost effectiveness ratio). Quality adjusted life years were estimated using a utility score ranging from 0 (death) to 1.0 (perfect health) derived from the HUI3 questionnaire, combined with the total length of follow-up time for each patient at baseline 12 months
Time Frame: 1 year after treatment initiation
Measure: Mean (Standard Deviation); unit: quality adjusted life years
Arm/Group | Standard Management | Fast Track
Number analyzed (Participants) | 75 | 80
quality adjusted life years | 0.587 (0.306) | 0.654 (0.289)

ADVERSE EVENTS:
Time Frame: Adverse event data were not collected
Description: All-cause mortality, serious and other (not including serious) adverse events were not monitored/assessed.
  Since we did not assess or monitor adverse events, we have reported the number at risk as "0" and also the number of patients experiencing an adverse event as "0".
Arm/Group | Standard Management | Fast Track
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-01-25): https://cdn.clinicaltrials.gov/large-docs/85/NCT02191085/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-16): https://cdn.clinicaltrials.gov/large-docs/85/NCT02191085/SAP_001.pdf